CLINICAL TRIAL: NCT00302172
Title: A Phase 1 Dose Escalation Study of ARQ 197 in Adult Patients With Metastatic Solid Tumors
Brief Title: ARQ 197 in Subjects With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: ArQule, ArQule, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-101
Record Dates: First submitted 2006-03-10; First posted 2006-03-14 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Cancer; Tumor
Keywords: Cancer; solid tumor; metastatic; primary tumor
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARQ 197 (Experimental)
  Interventions: Drug: ARQ 197

INTERVENTIONS:
Drug: ARQ 197 — Patients in this trial will receive ARQ 197 orally at dose levels specified for their respective dose cohorts. Dosing will begin at 20 mg/day (first cohort) and escalate until the RP2D or MTD is determined. Patients enrolled under a previous amendment will continue to receive ARQ 197 twice daily for 14 days followed by 7 days without therapy. Any patient enrolled under Amendment 3 will take ARQ 197 twice daily for 21 days where cycles will be repeated every three-weeks (21 days).
  Patients enrolled under Amendment 4 will receive dose of 360 mg bid (720 mg daily) continuously for 21 days, and cycle will be repeated every three weeks.
  All patients will remain on study until progression of disease, unacceptable toxicity, or another discontinuation criterion is met. In the case of toxicity, dose adjustment is permitted.

SUMMARY:
To determine the safety, tolerability and recommended Phase 2 dose (RP2D) of ARQ 197.

DETAILED DESCRIPTION:
To determine the safety, tolerability and recommended Phase 2 dose (RP2D) of ARQ 197 given orally. This is an open label, dose escalation study of ARQ 197 administered orally at a starting dose of 10 mg bid (20 mg/day).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent must be obtained and documented according to ICH GCP, the local regulatory requirements, and permission to use private health information in accordance with HIPPA prior to study-specific screening procedures
* A histologically or cytologically confirmed RCC or other c-Met expression tumors that is metastatic
* Patient must have available archival tumor tissue or accessible tumor that is safely amenable to tumor biopsy
* ≥ 18 years of age
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors
* Karnofsky performance status ≥ 70%
* Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last ARQ 197 dose
* Females of childbearing potential must have a negative serum pregnancy test
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × upper limit of normal (ULN) or ≤ 5.0 × ULN with metastatic liver disease.
* Hemoglobin (Hgb) ≥ 10 g/dl
* Total bilirubin ≤ 1.5 × ULN
* Creatinine ≤ 1.5 x ULN
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L

Exclusion Criteria:

* Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within four weeks of first dose
* Surgery within 4 weeks prior to first dose
* Known brain metastases
* Pregnant or breastfeeding
* Significant gastrointestinal disorder(s), in the opinion of the Principal Investigator, (e.g., Crohn's disease, ulcerative colitis, extensive gastric resection)
* Unable or unwilling to swallow ARQ 197 capsules twice daily
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements
* Bradycardia at baseline or known history of arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2006-01

PRIMARY OUTCOMES:
safety, tolerability | All patients will remain on study until progression of disease, unacceptable toxicity, or another discontinuation criterion is met

SECONDARY OUTCOMES:
To determine the pharmacokinetic profile of ARQ 197. | All patients will remain on study until progression of disease, unacceptable toxicity, or another discontinuation criterion is met
To determine the pharmacodynamics (i.e., identify biomarkers) of ARQ 197. | All patients will remain on study until progression of disease, unacceptable toxicity, or another discontinuation criterion is met
To assess the preliminary anti-tumor activity of ARQ 197. | All patients will remain on study until progression of disease, unacceptable toxicity, or another discontinuation criterion is met

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Premiere Oncology, Santa Monica, California
  - The Cleveland Clinic, Cleveland, Ohio
  - Mary Crowley Medical Research Center, Dallas, Texas